CLINICAL TRIAL: NCT05167708
Title: The Effect of Single and Repeated Micro-osteoperforation on the Maxillary First Molar Distalization: A Randomized Controlled Trial
Brief Title: Effects of Micro-osteoperforation on the Maxillary First Molar Distalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Alaa alkasaby, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A03120219
Record Dates: First submitted 2021-11-30; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Accretions; Teeth
MeSH Terms: conditions — Dental Deposits

STUDY DESIGN:
Intervention Model Description: single-center, prospective, single blinded, with 3 parallel arms, randomized clinical trial that had a 1:1:1 allocation.
Who Masked: Outcomes Assessor
Masking Description: single blinded, the assessor of the out comes did not participate in the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): the group underwent distalization, with no Micro-osteoperforation
- Single MOP (Experimental): the group underwent one time Micro-osteoperforation procedure
  Interventions: Procedure: Micro-osteoperforation
- repeated MOP (Experimental): the group underwent monthly Micro-osteoperforation procedure
  Interventions: Procedure: Micro-osteoperforation

INTERVENTIONS:
Procedure: Micro-osteoperforation — flapless small punctures in the bone at direction of tooth movement to accelerate the movement.
  Arms: Single MOP; repeated MOP

SUMMARY:
the study aimed to evaluate the effect of different types of Micro-osteoperforation on the rate of distal movement of maxillary first molars as a primary out come. Besides, it was aimed to study secondary effect on the first molars by evaluating root resorption, bone density, and level of the pain during performing the procedures.

DETAILED DESCRIPTION:
in the study, investigators tried to evaluate two methods to accelerate tooth movement by comparing them with control group. the first method was to apply one-time micro-osteoperforation. the second method was to apply the micro-osteoperforation repeatedly till reaching the end of the phase one treatment.

ELIGIBILITY:
Inclusion Criteria:

* Space deficiency in the upper arch > 5 mm, and < 8 mm.
* Non-extraction lower arch.
* Full upper dentition up to the second molars.
* Third molar present in both sides, not yet erupted.

Exclusion Criteria:

* Systemic disease or syndrome.
* Evidence of root resorption.
* Poor oral hygiene.
* Previous orthodontic treatment
* Evidence of bone loss.
* Active periodontal disease.
* Pregnant females.
* Presence of oral habits

Ages: 16 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — sexual hormones could affect the study outcomes. aiming to minimize the factors that might cause bias of the results.
Enrollment: 30 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
rate of maxillary first molar distal movement | through study completion, an average 1 year
  evaluation of the whole rate of distal movement of the first molar

SECONDARY OUTCOMES:
decrease in length of maxillary first molars in mm. | through study completion, an average 1 year
  the change in the lengths of roots of maxillary first molars in mm.
bone density | through study completion, an average 1 year
  bone density around the first molar
pain perception questionnaire | through study completion, an average 1 year
  evaluate the pain perception to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: yasser lotfy, professor, Study Chair — Mansoura University; marwaa shamaa, ph.D, Study Director — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt